CLINICAL TRIAL: NCT04963101
Title: Characteristics of Transcriptome Expression Profile of PBMCs in Patients With Ossification of the Posterior Longitudinal Ligament
Brief Title: RNA-seq Analysis of PBMC in Patients With OPLL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fifth Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Huading Lu, Director of orthopaedics, Fifth Affiliated Hospital, Sun Yat-Sen University
Other Study IDs: ZDWY.CSYGJWK.003
Record Dates: First submitted 2021-07-02; First posted 2021-07-15 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-07

CONDITIONS: OPLL; PBMCs; Transcriptome; Bioinformatics

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this study, we planned to identify transcriptome expression profiles (circRNAs, lncRNAs, and mRNAs) from peripheral blood mononuclear cells (PBMCs) of 30 patients with OPLL and 30 other non-OPLL patients by high-throughput sequencing.Sequence analysis was used to predict miRNAs that might bind circRNAs and lncRNAs.Through bioinformatics analysis, competitive endogenous RNAs (cerRNAs), as well as coexpression networks among circRNAs, lncRNAs, miRNAs, and mRNAs, were constructed to provide key molecules and signaling pathways associated with OPLL.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily participate in the clinical study and sign the informed consent;
2. All OPLL patients meet the diagnostic criteria set out in the JOA Clinical Practice Guidelines for Spinal Ligament Osification 2019;
3. Age ≥18, gender unlimited;
4. All non-OPLL patients and healthy volunteers have no serious diseases of the heart, lung, brain, liver, kidney and blood system, such as autoimmune diseases, tumors, psychosis, infectious diseases, etc., and have no bad habits or recent history of taking special drugs.

Exclusion Criteria:

1. Unable to sign the informed consent;
2. Patients who do not meet the inclusion criteria or diagnostic criteria;
3. <18 years old;
4. Women planning to become pregnant/lactating/pregnant;
5. Complicated with serious heart, lung, brain, liver, kidney, blood system diseases, such as autoimmune diseases, tumors, mental illness, infectious diseases, drug addiction and other bad addicts;Those who have recently taken special drugs;
6. Individuals who do not agree to donate peripheral blood or who are obviously uncomfortable with drawing blood.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: A total of 30 peripheral blood samples were enrolled in this study, including 15 cases in the OPLL disease group and 15 cases in the non-OPLL control group.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-06-25 (Actual); Primary Completion 2022-06-25 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
circRNA, lncRNA, mRNA | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Facility, Zhuhai, Guangdong, China